CLINICAL TRIAL: NCT01560442
Title: Pupillometry and Pain Thresholds Patients Substituted by Methadone and Buprenorphine.
Acronym: PUPIDOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CSAPA ANPAA 63 (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-0117
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Opiate Dependent; Previous Illicit Drug Use
Keywords: Analgesics, opioids; Opiate substitution treatment; Methadone; Buprenorphine; Hyperalgesia; Pupil; Pain; Psychophysics; previous illicit drug intake, under a substitution program
MeSH Terms: conditions — Hyperalgesia; Pain | interventions — Buprenorphine; Methadone

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- buprenorphine
  Interventions: Drug: Buprenorphine and Methadone Hydrochloride
- Methadone Hydrochloride
  Interventions: Drug: Buprenorphine and Methadone Hydrochloride

INTERVENTIONS:
Drug: Buprenorphine and Methadone Hydrochloride — To study the relation between pupillary diameter measured under scotopic conditions, and the pain thresholds measured at the time of peak and residual effect of methadone / buprenorphine in opiate-dependent patients following a substitution program.

SUMMARY:
The purpose is to study the relation between pupillary diameter measured under scotopic conditions, and the pain thresholds measured at the time of peak and residual effect of methadone/buprenorphine in opiate-dependent patients following a substitution program.

DETAILED DESCRIPTION:
Patients substituted since at least 3 months shall be included during a regular control visit.

Each session shall consist in

* check for toxics in urine sample;
* measurement of pupil diameter;
* measurement of mechanical punctuate pain threshold;
* measurement of mechanical bone pain threshold.

A first session shall be done at time of residual effect of the opiate. A second session shall be done at time of peak effect of the opiate.

ELIGIBILITY:
Inclusion Criteria:

* substitution treatment stable since at least 3 months
* capacity to understand the protocol
* likely to come to visits
* covered by French welfare

Exclusion Criteria:

* chronic pain
* concomitant acute pain
* pregnancy or breast feeding
* relevant mental disease
* peripheral neuropathy
* diabetes
* regular intake of ketamine
* neuroleptic concomitant treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Opiate dependent patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of the pupil diameter | 24 hours after the last dose of treatment

SECONDARY OUTCOMES:
- The mechanical punctuate pain threshold as measured by Electronical Von Frey | 24 hours after the last dose of treatment, 3 hours after the last dose of methadone and 1 hour ½ after the last dose of buprenorphine
- The mechanical pressure pain threshold measured by Algometer on the tibial bone | 24 hours after the last dose of treatment, 3 hours after the last dose of methadone and 1 hour ½ after the last dose of buprenorphine
- The pupil diameter measured in scotopic .conditions (via infrared camera) at the hypothetical peak effect of either methadone or buprenorphine. | 24 hours after the last dose of treatment, 3 hours after the last dose of methadone and 1 hour ½ after the last dose of buprenorphine
- The pupil diameter measured in photopic conditions (via infrared camera) at the hypothetical residual effect of either methadone or buprenorphine | 24 hours after the last dose of treatment, 3 hours after the last dose of methadone and 1 hour ½ after the last dose of buprenorphine

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AUTHIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France